CLINICAL TRIAL: NCT03361137
Title: A Phase IV, Multicenter, Single-Arm, Open-Label Study of Emicizumab Prophylaxis in Patients With Hemophilia A With or Without Inhibitors Undergoing Minor Surgical Procedures
Brief Title: Study of Emicizumab Prophylaxis in Participants With Hemophilia A With or Without Inhibitors Undergoing Minor Surgical Procedures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The Sponsor decided to terminate the study early for several reasons (low enrollment, limited variety of surgery types, and available scientific data).
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML39791
Record Dates: First submitted 2017-11-20; First posted 2017-12-04 (Actual); Results first posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — emicizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- PwHA With Inhibitors, Emicizumab: Surgery Not Performed Cohort (Experimental): This cohort included participants with Hemophilia A (PwHA) with inhibitors that were enrolled but did not have surgery. All participants received emicizumab via subcutaneous (SC) injection at a loading dose of 3 milligrams of medication per kilogram of body weight (mg/kg) once weekly for the first 4 weeks, followed by 1.5 mg/kg once weekly, or by any other approved maintenance regimen, as long as they continued to derive sufficient benefit. Participants must have received all loading doses prior to surgery and planned to continue emicizumab for a minimum of 1 month after surgery.
  Interventions: Drug: Emicizumab
- PwHA With Inhibitors, Emicizumab: CVAD Removal Cohort (Experimental): This cohort included participants with Hemophilia A (PwHA) with inhibitors that were enrolled and had surgery for central venous access device (CVAD) removal. All participants received emicizumab via subcutaneous (SC) injection at a loading dose of 3 milligrams of medication per kilogram of body weight (mg/kg) once weekly for the first 4 weeks, followed by 1.5 mg/kg once weekly, or by any other approved maintenance regimen, as long as they continued to derive sufficient benefit. Participants must have received all loading doses prior to surgery and planned to continue emicizumab for a minimum of 1 month after surgery.
  Interventions: Drug: Emicizumab
- PwHA With Inhibitors, Emicizumab: Simple Dental Extraction Cohort (Experimental): This cohort included participants with Hemophilia A (PwHA) with inhibitors that were enrolled and had surgery for simple dental extraction. All participants received emicizumab via subcutaneous (SC) injection at a loading dose of 3 milligrams of medication per kilogram of body weight (mg/kg) once weekly for the first 4 weeks, followed by 1.5 mg/kg once weekly, or by any other approved maintenance regimen, as long as they continued to derive sufficient benefit. Participants must have received all loading doses prior to surgery and planned to continue emicizumab for a minimum of 1 month after surgery.
  Interventions: Drug: Emicizumab
- PwHA Without Inhibitors, Emicizumab: CVAD Removal Cohort (Experimental): This cohort included participants with Hemophilia A (PwHA) without inhibitors that were enrolled and had surgery for central venous access device (CVAD) removal. All participants received emicizumab via subcutaneous (SC) injection at a loading dose of 3 milligrams of medication per kilogram of body weight (mg/kg) once weekly for the first 4 weeks, followed by 1.5 mg/kg once weekly, or by any other approved maintenance regimen, as long as they continued to derive sufficient benefit. Participants must have received all loading doses prior to surgery and planned to continue emicizumab for a minimum of 1 month after surgery.
  Interventions: Drug: Emicizumab
- PwHA Without Inhibitors, Emicizumab: Simple Dental Extraction Cohort (Experimental): This cohort included participants with Hemophilia A (PwHA) without inhibitors that were enrolled and had surgery for simple dental extraction. All participants received emicizumab via subcutaneous (SC) injection at a loading dose of 3 milligrams of medication per kilogram of body weight (mg/kg) once weekly for the first 4 weeks, followed by 1.5 mg/kg once weekly, or by any other approved maintenance regimen, as long as they continued to derive sufficient benefit. Participants must have received all loading doses prior to surgery and planned to continue emicizumab for a minimum of 1 month after surgery.
  Interventions: Drug: Emicizumab

INTERVENTIONS:
Drug: Emicizumab — Emicizumab via SC injection at a loading dose 3 mg/kg once weekly for the first 4 weeks, followed by 1.5 mg/kg once weekly, or by any other approved maintenance regimen, as long as the participant continues to derive sufficient benefit. Dosing was to be adjusted if the participant had a significant change in body weight.
  Other Names: Hemlibra®; ACE910; RG6013

SUMMARY:
This Phase IV, multicenter study will evaluate whether participants with Hemophilia A (PwHA) with or without inhibitors receiving emicizumab prophylaxis can safely undergo minor surgical procedures without additional prophylactic bypassing agents (BPA; for participants with inhibitors) or factor VIII (FVIII; for participants without inhibitors).

ELIGIBILITY:
Inclusion Criteria:

* Any age (newborn and older)
* Ability to comply with the study protocol, in the investigator's judgment
* Diagnosis of hemophilia A and current or history of an inhibitor (Bethesda titer ≥0.6 Bethesda units) and currently using bypassing agents (BPAs) for breakthrough bleeds (for PwHA with inhibitors)
* Diagnosis of hemophilia A and no history of an inhibitor (Bethesda titer <0.6 Bethesda units), or a history of an inhibitor that has been tolerized for >5 years and using FVIII for breakthrough bleeds (for PwHA without inhibitors)
* Plan to receive at least 4 loading doses of emicizumab and been adherent to emicizumab prophylaxis by the time of surgery
* Undergoing minor surgery within 60 days of study enrollment. Other minor surgical procedures could be included upon consultation and approval of Medical Monitor, but examples include central venous catheter insertion/removal/replacement, simple dental extractions, colonoscopy, cystoscopy, or endoscopy with biopsy, excisional skin biopsy
* Must plan to continue emicizumab prophylaxis for at least 1 month after surgery
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year during the study period

Exclusion Criteria:

* Diagnosis of a bleeding disorder other than hemophilia A
* Participants who have been tolerized to Factor VIII products (for PwHA with inhibitors)
* Tolerized to FVIII products for <5 years (for PwHA without inhibitors)
* Using FVIII products to treat breakthrough bleeds (for PwHA with inhibitors)
* Treatment with BPAs or FVIII within 24 hours prior to surgical procedure
* Undergoing a major surgical procedure
* Previous (in the past 12 months) or current treatment for thromboembolic disease (with the exception of previous catheter-associated thrombosis for which anti-thrombotic treatment is not currently ongoing) or current signs of thromboembolic disease
* Other conditions (e.g., certain autoimmune diseases, including but not limited to diseases such as systemic lupus erythematosus, inflammatory bowel disease, and antiphospholipid syndrome) that may increase the risk of bleeding or thrombosis
* Patients who are at high risk for thrombotic microangiopathy (TMA), e.g., have a previous medical or family history of TMA, in the investigator's judgment
* Would refuse treatment with blood or blood products, if necessary
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the participant's safe participation in and completion of the study
* Pregnant or lactating, or intending to become pregnant during the study; women of childbearing potential must have a negative serum pregnancy test result within 7 days before Study Day 1
* Treatment with any of the following: An investigational drug to treat or reduce the risk of hemophilic bleeds within 5 half-lives of last drug administration before Study Day 1; A non-hemophilia-related investigational drug within the last 30 days or 5 half-lives before Study Day 1 (whichever is longer); An investigational drug concurrently
* History of clinically significant hypersensitivity associated with monoclonal antibody therapies or components of the emicizumab injection
* Known human immunodeficiency virus (HIV) infection with CD4 count < 200 cells/microlitre within 24 weeks prior to enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- United States (8):
  - Childrens Hospital of LA, Los Angeles, California
  - Stanford University/Lucile Packard Children's Hospital, Palo Alto, California
  - University of Florida, Gainesville, Florida
  - Indiana Hemophilia & Thrombosis center, Indianapolis, Indiana
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - State University of New York at Buffalo; Women's and Children's Hospital of Buffalo, Buffalo, New York
  - Cook Childrens Medical Center, Fort Worth, Texas
  - University of Utah; Division of Gastroenterology/Hepatology, Salt Lake City, Utah

REFERENCES:
- [Background] Blanchette VS, Key NS, Ljung LR, Manco-Johnson MJ, van den Berg HM, Srivastava A; Subcommittee on Factor VIII, Factor IX and Rare Coagulation Disorders of the Scientific and Standardization Committee of the International Society on Thrombosis and Hemostasis. Definitions in hemophilia: communication from the SSC of the ISTH. J Thromb Haemost. 2014 Nov;12(11):1935-9. doi: 10.1111/jth.12672. Epub 2014 Sep 3. No abstract available. PMID 25059285

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PwHA With Inhibitors, Emicizumab: Surgery Not Performed Cohort | PwHA With Inhibitors, Emicizumab: CVAD Removal Cohort | PwHA With Inhibitors, Emicizumab: Simple Dental Extraction Cohort | PwHA Without Inhibitors, Emicizumab: CVAD Removal Cohort | PwHA Without Inhibitors, Emicizumab: Simple Dental Extraction Cohort
Started | 1 | 9 | 1 | 2 | 1
Completed | 0 | 9 | 1 | 2 | 1
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Reason not specified | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PwHA With Inhibitors, Emicizumab: Surgery Not Performed Cohort | PwHA With Inhibitors, Emicizumab: CVAD Removal Cohort | PwHA With Inhibitors, Emicizumab: Simple Dental Extraction Cohort | PwHA Without Inhibitors, Emicizumab: CVAD Removal Cohort | PwHA Without Inhibitors, Emicizumab: Simple Dental Extraction Cohort | Total
Number analyzed (Participants) | 1 | 9 | 1 | 2 | 1 | 14
Age, Customized [Count of Participants; unit: Participants]
  <18 Years Old | 1 | 7 | 1 | 2 | 0 | 11
  ≥18 to <65 Years Old | 0 | 2 | 0 | 0 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 1 | 9 | 1 | 2 | 1 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 1 | 1 | 0 | 5
  Not Hispanic or Latino | 1 | 6 | 0 | 1 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 1 | 0 | 0 | 0 | 1 | 2
  White | 0 | 5 | 1 | 1 | 0 | 7
  Multiple | 0 | 2 | 0 | 0 | 0 | 2
  Unknown | 0 | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Without Excessive Bleeding at Surgical Sites and Did Not Require BPA/FVIII Use for Bleeding Related to the Surgery, From the Start of Surgery Until Discharge, as Measured by the ISTH Hemostatic Efficacy Scale
Description: The International Society on Thrombosis and Haemostasis (ISTH) Assessment of Hemostatic Response for Surgical Procedures scale (see reference PubMed ID:25059285) has four categories, listed here in order of best to worst response: Excellent, Good, Fair, and Poor. The participant's bleeding related to surgery was evaluated by the healthcare professional who performed the procedure using the hemostatic efficacy scale, with an absence of excessive bleeding at the surgical site indicated by a good to excellent rating. The endpoint was met when the response to "Intraoperative and/or postoperative blood loss increased over expectation for the non-hemophilic patient determined at the time of discharge" was "0 to <10%" or "10% to < 25%" AND the response to the question "Did the patient use any bypassing agent (BPA)/factor VIII (FVIII) for the surgery before the discharge?" was "No".
Time Frame: Determined at the time of discharge (within approximately 48 hours after surgery)
Population: Efficacy Analysis Population: All enrolled participants who received emicizumab and underwent a minor surgery. One participant with hemophilia A with inhibitors did not undergo surgery and was therefore excluded from efficacy analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | PwHA With Inhibitors, Emicizumab: Surgery Not Performed Cohort | PwHA With Inhibitors, Emicizumab: CVAD Removal Cohort | PwHA With Inhibitors, Emicizumab: Simple Dental Extraction Cohort | PwHA Without Inhibitors, Emicizumab: CVAD Removal Cohort | PwHA Without Inhibitors, Emicizumab: Simple Dental Extraction Cohort
Number analyzed (Participants) | 0 | 9 | 1 | 2 | 1
Percentage of participants |  | 66.7 | 100.0 | 100.0 | 100.0

2. Primary Outcome: Percentage of Participants With Excessive Bleeding at Surgical Sites and Required BPA/FVIII Use for Treating Bleeding Related to the Surgery, From the Start of Surgery Until Discharge, as Measured by the ISTH Hemostatic Efficacy Scale
Description: The ISTH Assessment of Hemostatic Response for Surgical Procedures scale (see reference PubMed ID:25059285) has four categories, listed here in order of best to worst response: Excellent, Good, Fair, and Poor. The participant's bleeding related to surgery was evaluated by the healthcare professional who performed the procedure using the hemostatic efficacy scale, with excessive bleeding at the surgical site indicated by a fair to poor rating. The endpoint was met when the response to "Intraoperative and/or postoperative blood loss increased over expectation for the non-hemophilic patient determined at the time of discharge" was "25% to <50%" or "≥50%" AND the response to the question "Did the patient use any bypassing agent (BPA)/factor VIII (FVIII) for the surgery before the discharge?" was "Yes". The percentage of participants by type and dose of BPA/FVIII used to treat the bleeding is also reported. rFVIIa = recombinant activated human factor VII (eptacog alfa [activated])
Time Frame: Determined at the time of discharge (within approximately 48 hours after surgery)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | PwHA With Inhibitors, Emicizumab: Surgery Not Performed Cohort | PwHA With Inhibitors, Emicizumab: CVAD Removal Cohort | PwHA With Inhibitors, Emicizumab: Simple Dental Extraction Cohort | PwHA Without Inhibitors, Emicizumab: CVAD Removal Cohort | PwHA Without Inhibitors, Emicizumab: Simple Dental Extraction Cohort
Number analyzed (Participants) | 0 | 9 | 1 | 2 | 1
Percentage of participants
  Total with Excessive Bleeding and Received BPA/FVIII |  | 11.1 | 0.0 | 0.0 | 0.0
  Treated with 2 mg rFVIIa |  | 11.1 | 0.0 | 0.0 | 0.0

3. Primary Outcome: Percentage of Participants Who, After Being Discharged From Surgery, Experienced Bleeds That Were Either Related or Unrelated to Surgery and Also Required BPA/FVIII Use
Description: Post-surgical bleeding information was self-reported by participants (or the participant's legally authorized representative) on the "Bleed and Medication Diary". Bypassing agents (BPAs)/factor VIII (FVIII) used to treat excessive bleeding were also self-reported by participants if it was self-administered. BPAs/FVIII administered by the investigators to treat the bleeding were reported on the "Concomitant Medications" case report form page. The percentage of participants by type and dose of BPA/FVIII used to treat the bleeding is also reported. rFVIIa = recombinant activated human factor VII (eptacog alfa [activated])
Time Frame: Within 48 hours (if discharged home), and 8 and 28 days after surgery
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | PwHA With Inhibitors, Emicizumab: Surgery Not Performed Cohort | PwHA With Inhibitors, Emicizumab: CVAD Removal Cohort | PwHA With Inhibitors, Emicizumab: Simple Dental Extraction Cohort | PwHA Without Inhibitors, Emicizumab: CVAD Removal Cohort | PwHA Without Inhibitors, Emicizumab: Simple Dental Extraction Cohort
Number analyzed (Participants) | 0 | 9 | 1 | 2 | 1
Percentage of participants
  Total with Post-surgical Bleeding and Received BPA/FVIII |  | 22.2 | 100.0 | 0.0 | 0.0
  Treated with 2 mg rFVIIa |  | 11.1 | 100.0 | 0.0 | 0.0
  Treated with 5 mg rFVIIa |  | 11.1 | 0.0 | 0.0 | 0.0

4. Primary Outcome: Emicizumab Plasma Concentration on the Day of Surgery
Description: Enrolled participants received a minimum of four loading doses of emicizumab prior to their surgical procedure. Pharmacokinetic blood samples were obtained at study sites 24 hours before the procedures in order to describe emicizumab plasma concentration on the day of surgery for each of the inhibitor and non-inhibitor cohorts.
Time Frame: Approximately 24 hours prior to surgery
Population: Efficacy Analysis Population: All enrolled participants who received emicizumab and underwent a minor surgery. One participant with hemophilia A with inhibitors did not undergo surgery and was therefore excluded from this analysis.
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (μg/mL)
Groups:
- PwHA With Inhibitors, Emicizumab: All Surgery Cohorts: This analysis set included all participants with Hemophilia A (PwHA) with inhibitors who had undergone surgery. All participants received emicizumab via subcutaneous (SC) injection at a loading dose of 3 milligrams of medication per kilogram of body weight (mg/kg) once weekly for the first 4 weeks, followed by 1.5 mg/kg once weekly, or by any other approved maintenance regimen, as long as they continued to derive sufficient benefit. Participants must have received all loading doses prior to surgery and planned to continue emicizumab for a minimum of 1 month after surgery.
- PwHA Without Inhibitors, Emicizumab: All Surgery Cohorts: This analysis set included all participants with Hemophilia A (PwHA) without inhibitors who had undergone surgery. All participants received emicizumab via subcutaneous (SC) injection at a loading dose of 3 milligrams of medication per kilogram of body weight (mg/kg) once weekly for the first 4 weeks, followed by 1.5 mg/kg once weekly, or by any other approved maintenance regimen, as long as they continued to derive sufficient benefit. Participants must have received all loading doses prior to surgery and planned to continue emicizumab for a minimum of 1 month after surgery.
Arm/Group | PwHA With Inhibitors, Emicizumab: All Surgery Cohorts | PwHA Without Inhibitors, Emicizumab: All Surgery Cohorts
Number analyzed (Participants) | 10 | 3
micrograms per millilitre (μg/mL) | 53.74 (28.67) | 38.40 (8.95)

5. Primary Outcome: Safety Summary of the Number of Participants With at Least One Adverse Event
Description: All adverse events (AEs) that occurred after informed consent was obtained were coded using the Medical Dictionary for Regulatory Activities (MedDRA) v23.0, summarized by severity according to the World Health Organization (WHO) toxicity grading scale (Grade 1 is mild; Grade 2 is moderate; Grade 3 is severe; Grade 4 is life-threatening; and Grade 5 is death related to AE), and tabulated by body system and preferred term (PT) for individual events within each system organ class (SOC). For each AE, the investigator independently assessed its severity and seriousness, and whether it was considered to be related to the study drug.
Time Frame: From Baseline up to 30 days after surgery
Population: The analysis included all enrolled participants who provided informed consent.
Measure: Count of Participants; unit: Participants
Arm/Group | PwHA With Inhibitors, Emicizumab: Surgery Not Performed Cohort | PwHA With Inhibitors, Emicizumab: CVAD Removal Cohort | PwHA With Inhibitors, Emicizumab: Simple Dental Extraction Cohort | PwHA Without Inhibitors, Emicizumab: CVAD Removal Cohort | PwHA Without Inhibitors, Emicizumab: Simple Dental Extraction Cohort
Number analyzed (Participants) | 1 | 9 | 1 | 2 | 1
Participants
  Any Adverse Event (AE) | 1 | 4 | 0 | 0 | 0
  AE with Fatal Outcome | 0 | 0 | 0 | 0 | 0
  Serious Adverse Event (SAE) | 0 | 0 | 0 | 0 | 0
  SAE Leading to Withdrawal from Treatment | 0 | 0 | 0 | 0 | 0
  SAE Leading to Dose Modification/Interruption | 0 | 0 | 0 | 0 | 0
  Related SAE | 0 | 0 | 0 | 0 | 0
  AE Leading to Withdrawal from Treatment | 0 | 0 | 0 | 0 | 0
  AE Leading to Dose Modification/Interruption | 0 | 0 | 0 | 0 | 0
  Related AE | 0 | 0 | 0 | 0 | 0
  Related AE Leading to Withdrawal from Treatment | 0 | 0 | 0 | 0 | 0
  Related AE Leading to Dose Modification/Interruption | 0 | 0 | 0 | 0 | 0
  Grade 3-5 AE | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Percentage of Participants With Surgical Complications Requiring Hospitalization or Return to Surgery
Description: This safety endpoint was a composite endpoint. Surgical complications were entered as adverse events on the case report form page with "Other suspected causes" marked as "Study Surgery or Procedure". This endpoint was met when response to "It required or prolonged inpatient hospitalization" was checked OR response to "Was procedure/surgery performed?" was "Yes".
Time Frame: Within 48 hours after surgery, and 8 and 28 days after initial surgery
Population: The analysis included all enrolled participants who received emicizumab and underwent a minor surgery. One participant with hemophilia A with inhibitors did not undergo surgery and was therefore excluded from analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | PwHA With Inhibitors, Emicizumab: Surgery Not Performed Cohort | PwHA With Inhibitors, Emicizumab: CVAD Removal Cohort | PwHA With Inhibitors, Emicizumab: Simple Dental Extraction Cohort | PwHA Without Inhibitors, Emicizumab: CVAD Removal Cohort | PwHA Without Inhibitors, Emicizumab: Simple Dental Extraction Cohort
Number analyzed (Participants) | 0 | 9 | 1 | 2 | 1
Percentage of participants |  | 0.0 | 0.0 | 0.0 | 0.0

7. Primary Outcome: Percentage of Participants Who Needed Blood/Blood Product Transfusions During Surgery
Description: The percentage of participants who needed blood or blood product transfusions (e.g., platelets, plasma, etc.) during surgery was evaluated.
Time Frame: Within 48 hours after surgery, and 8 and 28 days after initial surgery
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | PwHA With Inhibitors, Emicizumab: Surgery Not Performed Cohort | PwHA With Inhibitors, Emicizumab: CVAD Removal Cohort | PwHA With Inhibitors, Emicizumab: Simple Dental Extraction Cohort | PwHA Without Inhibitors, Emicizumab: CVAD Removal Cohort | PwHA Without Inhibitors, Emicizumab: Simple Dental Extraction Cohort
Number analyzed (Participants) | 0 | 9 | 1 | 2 | 1
Percentage of participants |  | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: From Baseline up to 30 days after surgery
Arm/Group | PwHA With Inhibitors, Emicizumab: Surgery Not Performed Cohort | PwHA With Inhibitors, Emicizumab: CVAD Removal Cohort | PwHA With Inhibitors, Emicizumab: Simple Dental Extraction Cohort | PwHA Without Inhibitors, Emicizumab: CVAD Removal Cohort | PwHA Without Inhibitors, Emicizumab: Simple Dental Extraction Cohort
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/9 | 0/1 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/9 | 0/1 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 4/9 | 0/1 | 0/2 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PwHA With Inhibitors, Emicizumab: Surgery Not Performed Cohort (N=1) | PwHA With Inhibitors, Emicizumab: CVAD Removal Cohort (N=9) | PwHA With Inhibitors, Emicizumab: Simple Dental Extraction Cohort (N=1) | PwHA Without Inhibitors, Emicizumab: CVAD Removal Cohort (N=2) | PwHA Without Inhibitors, Emicizumab: Simple Dental Extraction Cohort (N=1)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adhesiolysis (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
No definitive efficacy conclusions were drawn due to study limitations that included early enrollment termination, limited number of participants enrolled, and evaluation in only 2 minor surgical procedure types.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but only after the first publication or presentation that involves the overall study. The Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT03361137/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/37/NCT03361137/SAP_001.pdf